CLINICAL TRIAL: NCT05007405
Title: Spectrum of Bacterial Infections in Rheumatology and the Role of Urinary Tract Infection
Brief Title: Spectrum of Bacterial Infections in Rheumatology
Acronym: SIBERIE
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD 1820
Record Dates: First submitted 2021-08-11; First posted 2021-08-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-08

CONDITIONS: Articular Disease
Keywords: Osteoarticular infection; Bacteria; Urinary tract infections
MeSH Terms: conditions — Joint Diseases; Urinary Tract Infections | interventions — Population Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Osteoarticular infections: Retrospective study on medical file of patients with osteoarticular infections diagnose (date of the positive bacteriological sample) between January 1, 2010 and December 31, 2020
  Interventions: Other: Groups/Cohortes

INTERVENTIONS:
Other: Groups/Cohortes — Retrospective study on medical file of patients with osteoarticular infections diagnose (date of the positive bacteriological sample) between January 1, 2010 and December 31, 2020
  Other Names: Osteoarticular infections

SUMMARY:
Retrospective study of patients with a proved non-tuberculous osteoarticular infection (OAI) diagnosed in a rheumatology department during the years 2010-2020. The objectives are :

* To describe sites, type of micro-organism, clinical data, origin of infection, therapeutic modalities et outcome
* To compare OAI of urinary origin with those with another origin

DETAILED DESCRIPTION:
This retrospective study will be conducted on medical files. Patients will be mainly selected on :

* A proved osteoarticular infection (OAI) diagnosed in the department of rheumatology of the René Dubos hospital from 1° January 2010 to 31 December 2020.
* Adult patients 18 year's old or older
* Infection proved by positive culture in the osteoarticular site and/or blood (with typical clinical and imaging features)

The followed OAI are not included :

* Infection on prosthetic joint, materiel ; post-operative OAI ; osteomyelitis
* Brucellosis ; Lyme disease

Patients are selected from the codification of the hospitalization ; medical files are reviewed by the investigators.

OAI of urinary origin is defined either by the same micro-organism in urine and osteo-articular sample (or blood) or a bacteria in the osteo-articular sample in conjunction with : urologic pathology, recurrent urinary tract infection, urologic surgery, antibiotic therapy.

* Characteristics of three populations will be compared :
* - OAI of urinary origin
* - OAI of another origin (skin, etc)
* - OAI without known origin Characteristics include : gender, age, risk factors, site of osteo-articular infection, type of micro-organism, type of positive sample(s), blood cultures, urinary cultures, duration of symptoms, site of primary infection and/or type of contamination, biological results, echocardiography, imaging results, type of treatment (medical, surgical), outcome, duration of hospitalization, intensive unit care stay, death at hospital.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 years and over at the time of diagnosis
* Osteoarticular infection (septic arthritis, spondylodiscitis), by a bacterium or a fungus, proven by a bacteriological sample in situ or in the blood by positive blood culture (with an unequivocal clinical, biological and imaging feature),
* Diagnosed between 01/01/2010 and 12/31/2020 (11 years)
* Hospitalization in the rheumatology department of CH René Dubos, Pontoise

Exclusion Criteria:

* Bacterial infection due to the following germs: mycobacteria, brucella, Borrelia
* Early infection on joint prosthesis
* Peripheral osteomyelitis
* Osteoarticular infection without bacteriological proof

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarticular infections diagnose (date of the positive bacteriological sample) between January 1, 2010 and December 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of the spectrum of osteoarticular infections in adult, in a rheumatology department | Through study completion, an average of 1 year
  The purpose of this database is to describe the spectrum of osteoarticular infections in adults, non-tuberculosis germs, in a rheumatology department of a CHG during the 2010s

SECONDARY OUTCOMES:
Prevalence of urinary origin in osteoarticular infections in adults, compared with other origins | Through study completion, an average of 1 year
  The second purpose of this database is to identify the characteristics of osteo-articular infections of urinary origin

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Pertuiset, Dr, Principal Investigator — Hôpital NOVO
Locations (1):
- Department of Rheumatology, Hospital René Dubos, Pontoise, Pontoise, France

REFERENCES:
- [Background] Ross JJ. Septic Arthritis of Native Joints. Infect Dis Clin North Am. 2017 Jun;31(2):203-218. doi: 10.1016/j.idc.2017.01.001. Epub 2017 Mar 30. PMID 28366221
- [Background] Berbari EF, Kanj SS, Kowalski TJ, Darouiche RO, Widmer AF, Schmitt SK, Hendershot EF, Holtom PD, Huddleston PM 3rd, Petermann GW, Osmon DR, Infectious Diseases Society of America. 2015 Infectious Diseases Society of America (IDSA) Clinical Practice Guidelines for the Diagnosis and Treatment of Native Vertebral Osteomyelitis in Adults. Clin Infect Dis. 2015 Sep 15;61(6):e26-46. doi: 10.1093/cid/civ482. Epub 2015 Jul 29. PMID 26229122